CLINICAL TRIAL: NCT01251705
Title: Comparation of Different Devices to Measure Corneal Thickness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: L.E. Pillunat, University of Dresden
Other Study IDs: CompCornea
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Corneal Thickness
Keywords: Cornea; SL OCT; Spectral OCT Cornea modul; ultrasound pachymetry; Pentacam
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of different methods for measuring peoples corneal thickness

DETAILED DESCRIPTION:
Volunteers with healthy corneas will be measured by different instruments to detect their corneal thickness. First interindividual difference between the instruments will be reviewed. People will be measured again two times on two different days to examine an interindividual difference in all instruments.

ELIGIBILITY:
Inclusion Criteria:

* healthy cornea

Exclusion Criteria:

* myopia or astigmatism over 1,5 dpt
* corneal surgery
* acute ocular inflammation
* lost of vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteers without corneal disease
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Haustein, Doctor med., Principal Investigator — Departement of Ophthalmology University of Dresden
Locations (1):
- Departement of Ophthalmology, Dresden, Saxony, Germany